CLINICAL TRIAL: NCT02262247
Title: A Multicenter OUS Post-Market Clinical Follow-Up of the Medrobotics Flex® Robotic System Used for Accessing and Visualizing the Oropharynx, Hypopharynx, and Larynx During Transoral Procedures
Brief Title: A Post-Market Clinical Trial for Access and Visualization of the Oropharynx, Hypopharynx and Larynx During Transoral Procedures
Status: Completed | Type: Observational
Sponsor: Medrobotics Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: FLX-ENT-PMK-OUS-001
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: OSA; Oral Disease; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms
Keywords: Transoral; Oropharynx; Hypopharynx; Endoscopic; TORS; Endoscopic Transoral; Larynx
MeSH Terms: conditions — Mouth Diseases; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transoral Visualization & Access: Subjects ≥ 22 yrs requiring transoral procedures

SUMMARY:
The objectives of this study are to evaluate the performance of the Medrobotics Flex® Robotic System to visualize and access specific anatomical locations along with evaluation of the safety of the device.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 22 years of age
* Candidate for transoral surgery in the oropharynx, hypopharynx and larynx

Exclusion Criteria:

* Less than 22 years of age
* Not a candidate for transoral surgery in the oropharynx, hypopharynx and larynx

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 22 years of age requiring transoral procedures
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Access and Visualizaton in Oropharynx, Hypopharynx and Larynx | Intra-Operative
  Ability to access and visualize all the following anatomical locations in the oropharynx, hypopharynx and larynx via transoral only approach. Palatine tonsils, base of tongue, epiglottis, posterior pharyngeal wall, false vocal cords.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Tricoli, BS, MBA, Study Director — Medrobotics Corp
Locations (4):
- University Hospital of Louvain at Mont-Godinne, Yvoir, Belgium
- Germany (3):
  - University Hospital Ulm, Ulm, Baden-Wurttemberg
  - University Hosptial Giessen and Marburg, Marburg, Baldingerstraße
  - University Hospital of Essen, Essen, Hufelandstraße

IPD SHARING:
Plan to Share IPD: No